CLINICAL TRIAL: NCT00199147
Title: Treatment of Elderly Patients (>60 Years) With Acute Myeloblastic Leukemia or Advanced MDS (RAEB-T): An Open Randomized Study to Test the Efficacy of G-CSF-Priming and a Feasibility Trial of Dose-Reduced Allogeneic Transplantation and of Autologous Stem Cell Transplantation
Brief Title: Efficacy of G-CSF-Priming in Elderly AML Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML-elderly 01/99 Trial
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2005-10-26 (Estimated); Status verified 2005-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Etoposide; Idarubicin; Granulocyte Colony-Stimulating Factor; fludarabine; Stem Cell Transplantation

INTERVENTIONS:
Drug: Cytarabine
Drug: Etoposide
Drug: Idarubicin
Drug: G-CSF
Drug: Fludarabine
Procedure: Stem cell apheresis
Procedure: Stem cell transplantation

SUMMARY:
Aim of the study is to compare the efficacy of intensive induction therapy with Cytarabine, Idarubicin and Etoposide (IdAV) given in parallel with (G-CSF priming) and followed by G-CSF versus the same IdAV chemotherapy only followed by G-CSF (without priming) in elderly patients with de novo AML, secondary AML and advanced MDS. Moreover, the ability to mobilize sufficient numbers of peripheral blood stem cells (PBSC) for autologous PBSC transplantation after consolidation therapy with dose-reduced FLAG-Ida chemotherapy followed by G-CSF will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of de-novo AML, FAB M0, 1, 2, 4-7 or
* Diagnosis of secondary AML after previous chemotherapy and/or radiation therapy or after preceeding MDS or
* Diagnosis of an advanced MDS, i.e. RAEB-t according to the FAB classification or
* Extramedullary AML (chloroma, "granulocytic sarcoma")
* Age greater than 60 years (not including 60 years)
* ECOG performance status 0, 1, or 2
* Written informed consent

Exclusion Criteria:

* Patients with a t(15;17) translocation
* Patients with severe cardiac disease (e.g. cardiac failure NYHA III/IV, myocardial infarction within the last 6 months; severe ventricular arrythmias (Lown III or IV)
* Patients with severe complications of the leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock.
* Severe pulmonary disease (diffusion capacity for CO2 of less than 50%)
* Significant renal dysfunction (creatinine clearance < 60/min/min)
* Bilirubin > 2mg% (>34.2 mmol/l)
* Patients with a clinically active second malignancy
* Patients with a psychiatric, addictive, or any disorder wich compromises ability to give truly informed consent for participating in this study
* HIV positivity
* Known refractoriness to platelet transfusion, inability to adequately substitute blood products

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2000-01

PRIMARY OUTCOMES:
-Remission rate after induction therapy
-Remission duration
-Disease free survival
-Overall survival

SECONDARY OUTCOMES:
-Toxicity according to WHO
-Death in induction therapy
-Feasibility to mobilize peripheral blood stem cells
-Feasibility to perform autologous or allogeneic stem cell transplantation in elderly patients

CONTACTS AND LOCATIONS:
Overall Officials: Oliver G Ottmann, MD, Study Chair — University Hospital, Medical Department II, Frankfurt, Germany
Locations (1):
- University Hospital, Medical Department II, Frankfurt, Germany